CLINICAL TRIAL: NCT02187276
Title: The Predictive Factors of Good Clinical Response to Cholinesterase Inhibitors in Mild and Moderate Alzheimer Disease and Mixed Dementia: a Naturalistic Study
Brief Title: The Predictive Factors of Good Clinical Response to Cholinesterase Inhibitors in Alzheimer Disease and Mixed Dementia
Status: Completed | Type: Observational
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Luís Felipe José Ravic de Miranda, Physician, Geriatrician, PhD Student, Federal University of Minas Gerais
Other Study IDs: 0172/2010
Record Dates: First submitted 2014-07-05; First posted 2014-07-11 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Alzheimer Disease, Late Onset
Keywords: Predictive factors of response; mild and moderate; Alzheimer disease; mixed dementia; APOE; polymorphisms of CYP 2D6
MeSH Terms: conditions — Alzheimer Disease; Lymphoma, Follicular; Mixed Dementias | interventions — Cholinesterase Inhibitors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Genetic and biochemical analyzes A blood sample (5 mL) was withdrawn from all patients on the first consultation for DNA extraction and APOE genotyping in its different allelic forms (Ɛ2, Ɛ3, Ɛ4). An additional blood sample (10 mL) was withdrawn from patients who took donepezil (51 patients) and was kept in a tube with heparin and frozen at - 70 ° C. In this group of patients, we genotyped the APOE and assessed the polymorphism of CYP 2D6 (*3,*4,*5,*6 and*10). This procedure was done when they came at 3, 6 and 12 months consultation, respectively.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Alzheimer disease or mixed dementia: Patients were evaluated four times. In the first consultation, without taking cholinesterase inhibitors (ChEI), after three, six and 12 months taking ChEI.
  Interventions: Drug: cholinesterase inhibitors

INTERVENTIONS:
Drug: cholinesterase inhibitors — The first group received donepezil (5 or 10 mg) the second group received galantamine (16 or 24 mg) The third group received rivastigmine (3 or 4,5 or 6 mg BID) according to the treating physician.
  Other Names: No applicable

SUMMARY:
Background and objectives: The aims of this naturalistic study were: to analyze factors which could be predictive of good response to cholinesterase inhibitors (ChEI), such as: age, sex, schooling, mild (CDR 1) or moderate Alzheimer's disease (AD),(CDR 2), Apoliprotein epsilon 4 (APOE Ɛ4), among others, in their cognitive and clinical response. We also classified patients according to their response to Mini mental State of Examination (MMSE). Finally we saw the polymorphisms of APO E and cytochrome P450 2D6 (CYP2D6) and tried to correlate the response with different allelic forms of Apo E and among others with wild type homozygotes (wt/wt) and their polymorphisms (CYP2D6*3,*4, *5, *6 and 10) of CYP 2D6.

Patients and Methods: 129 patients were diagnosed as AD or AD+cerebrovascular disease (CVD) mild or moderate. After 12 month-treatment, 97 patients completed the study. They were assessed (four) times. In the first visit, without taking ChEI, after 3, 6 and 12 month-treatment, they were taking donepezil or rivastigmine or galantamine. We also extracted 5 mL of blood sample to genotype the DNA. In each visit, we applied cognitive, functional, mood and behavior scales. Good responders were defined as those who scored > 2 in MMSE.

Results and Conclusion: In longitudinal analysis, patients with mild AD and good responders at 3 months were considered good responders at 12 months. We obtained a higher rate of good responders comparing with other researches (27.8%). There was no correlation between dose, APOE and CYP 2D6 polymorphisms, although we already obtained clinical results with the dose dosage of 5mg.

DETAILED DESCRIPTION:
Genomic DNA for genotyping was extracted from total blood samples collected in ethylenediaminetetraacetic acid (EDTA) (Wizard Genomic DNA Purification Kit: Promega®, USA) and kept frozen at seventy degrees Celsius negative (-70ºC) until analysis. For APOE genotyping (alleles Ɛ2, Ɛ3 and Ɛ4), DNA samples were amplified by polymerase chain reaction (PCR), followed by digestion with Haemophilus haemolyticus restriction endonuclease I (HhaI) and restriction fragment length polymorphism (RFLP) analysis, as previously described by Hixson and Vernier.

The CYP2D6*3, CYP2D6*4 and CYP2D6*6 alleles were investigated by tetra-primer PCR and the CYP2D6*5 allele, which presents the entire CYP2D6 gene deletion, was identified by long PCR reaction, according to the method described by Hersberger et al. The CYP2D6*10 allele was amplified by PCR following Baclig et al. and the RFLP analysis was performed with Type II restriction enzyme (HphI). For all analysis a positive and negative controls were included.

Subjects carrying Epsilon 3, Epsilon 3 (Ɛ3Ɛ3), CYP2D6*3/4/5/6/10-nor specific mutations are classified as wild-type and functional allele carriers. The subjects carrying two defective alleles were classified as poor metabolizers (PM) and those heterozygous were classified as extensive metabolizers (EM).

ELIGIBILITY:
Inclusion Criteria:

- AD diagnosis or AD with CVD according the criteria of National Institute on Aging and the Alzheimer's Association workgroup and the National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA)

Exclusion Criteria:

* Patients with mild cognitive impairment;
* Other types of dementia, such as pure vascular dementia, frontotemporal dementia, dementia with Lewy bodies, corticobasal degeneration;
* Severe dementia (CDR 3)
* Those who were already taking ChEI,
* If there have not been agreement between the first researcher and the treating physician.

Ages: 59 Years to 92 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients were those who spontaneously went to the outpatient units to be diagnosed and presented cognitive, functional, and in many cases, behavioral symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2009-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Cognitive results | Patients were evaluated from 06/2009 to 03/2013 for four times - first visit ( without taking medication), after three, six and 12 months of treatment with cholinesterase inhibitors (up to 12 months)
  Clinical assessment: The clinical domains examined and the respective evaluation tools were: global cognition - MMSE, clock drawing test score and Mattis Dementia Rating Scale - DRS). Patients were seen between 06/2009 to 03/2013. Good clinical responders were those who scored ≥ 2 on the MMSE after 12 month-treatment, the neutrals had the scores between -1 and +1, and bad responders scored ≤ -2 at the same period. A subgroup who scored > 2 on the MMSE were defined as very good responders. Patients were seen for four times: at the first consultation (n=129), at three (n=114), six (n=105) and twelve months of treatment (n=97).

SECONDARY OUTCOMES:
Genetic and biochemical analyzes | To correlate allelic forms of APOE and CYP 2D6 polymorphisms with the response (up to 12 months)
  Genomic DNA for genotyping was extracted from total blood samples collected in EDTA (Wizard Genomic DNA Purification Kit: Promega®, USA) and kept frozen at -70ºC until analysis. For APOE genotyping (alleles Ɛ2, Ɛ3 and Ɛ4), DNA samples were amplified by polymerase chain reaction (PCR), followed by digestion with HhaI and restriction fragment length polymorphism (RFLP) analysis, as previously described by Subjects carrying Ɛ3Ɛ3, CYP2D6*3/4/5/6/10-nor specific mutations are classified as wild-type and functional allele carriers.Patients were seen four times (see Primary outcome).

OTHER OUTCOMES:
Determination of the concentration of donepezil | After 12 months-treatment the concentration of donepezil was measured
  We used Liquid chromatography-electrospray ionization tandem mass spectrometry for the quantitation of donepezil concentration in human plasma which was 05-250ng/mL.
  The analyses were carried out on a Waters system, composed of a 1525 binary pump, a 2777 sample manager, a TCM/CHM column oven and a Quattro LC triple quadrupole mass spectrometer, equipped with an electrospray ion source used in the positive ionization mode. MassLynx v.4.1 software was used for analysis. LC separation was performed on an ACE C18 column from ACT, at 30 ◦C. The mobile phase consisted of 2 mM aqueous ammonium acetate (pH 3.2) adjusted with formic acid and methanol (38:62), at a flow rate of 1 mL/min. The run time was 2.8 min and the injection volume was 20 µL. Internal standard is Indapamida. Analytes were extracted from plasma samples by a protein precipitation procedure using methanol. The method was developed and validated according the FDA guidance for bioavailability and bioequivalence studies.

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Caramelli, Profesor, Study Chair — Federal University of Minas Gerais